CLINICAL TRIAL: NCT02913404
Title: Functional Biomechanical Outcome of ACL-reconstruction vs. ACL-reconstruction and Extra-articular-tenodesis in Patients
Brief Title: ACL-reconstruction vs ACL-reconstruction With EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, William Anderst, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO16080675
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: ACL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL Reconstruction (Experimental): Surgical Protocol
  Standard single bundle anatomic ACL reconstruction will be performed for all subjects. Quadrupled hamstring tendon will be used with cortical fixation on femur and tibia.
  Interventions: Procedure: ACL Reconstruction
- ACL Recon. extra-articular-tenodesis (Experimental): Surgical Protocol
  Standard single bundle anatomic ACL reconstruction will be performed for all subjects. Quadrupled hamstring tendon will be used with cortical fixation on femur and tibia. ACL-R+EAT will be performed as described by Marcacci with doubled hamstring tendon left attached at the pes anserinus, an anatomic tibial tunnel, staple fixation in the over the top position, routing of the graft superficial to the LCL, and staple fixation at Gerdy's tubercle. Concomitant tears to the menisci and their roots will be repaired as indicated.
  Interventions: Procedure: ACL Recon. extra-articular-tenodesis

INTERVENTIONS:
Procedure: ACL Reconstruction — standard surgical procedure
  Arms: ACL Reconstruction
Procedure: ACL Recon. extra-articular-tenodesis — standard surgical procedure and extra-articular-tenodesis will be used for a randomized portion of participants
  Arms: ACL Recon. extra-articular-tenodesis

SUMMARY:
The purpose of this study is to asses functional biomechanical outcomes and patient reported outcome measures following single bundle ACL reconstruction (ACL-R) compared to single bundle ACL reconstruction and extra articular tenodesis (ACL-R+EAT).

DETAILED DESCRIPTION:
Screening Protocol All participants that express interest in the study will receive a screening interview that will determine eligibility for participation in the study. The screening of surgical patients will be performed by one of the clinical research coordinators in the clinic of Dr. Musahl.

Potential participants who pass the screening interview will be provided a copy of the informed consent form (in person or via email). The potential participant will review the consent form in detail with a member of the clinical team in order to ensure that the participant understands the information contained in the consent form and to provide an opportunity for the participant to ask questions about the study. If the potential participant then agrees to participate, the consent form will be signed by the participant and a member of the clinical team.

Surgical Protocol Baseline testing before surgery will consist of the IKDC objective and subjective score, KOOS score, Marx activity level, Lysohm Scale and VR-12. A radiologist will grade clinical MRI for ACL, meniscus, MCL, LCL, and ALC injury. Quantitative pivot shift testing will be performed under anesthesia using the PIVOT technology and inertial sensor. Intraoperative grading of ACL injury and concomitant injuries to the articular cartilage and meniscus will be performed. If deemed eligible final randomization will occur following intraoperative grading.

Standard single bundle anatomic ACL reconstruction will be performed for all subjects. Quadrupled hamstring tendon will be used with cortical fixation on femur and tibia. ACL-R+EAT will be performed as described by Marcacci with doubled hamstring tendon left attached at the pes anserinus, an anatomic tibial tunnel, staple fixation in the over the top position, routing of the graft superficial to the LCL, and staple fixation at Gerdy's tubercle. Concomitant tears to the menisci and their roots will be repaired as indicated.

Research Scans After surgery, approximately 6 months, subjects will undergo a CT scan on bilateral knees. The CT scan will be used to create volumetric models. These bone models will be matched to the dynamic biplane x-rays. Subjects will also undergo a research MRI scan on bilateral knees. The MRI scan will be used to generate models of the knee articular cartilage.

Testing Protocol Participants who pass the screening interview, consent to participate in this study and undergo surgical treatment will be scheduled for two test sessions at the University of Pittsburgh Biodynamics Lab, a research CT scan and MRI scan at UPMC Presbyterian. The participant will then be assigned a study ID number that will be used to identify all de-identified data associated with the participant. The study ID number will be recorded and placed with the consent form in a folder that will remain in a locked file cabinet in the Biodynamics Lab.

Female participants will complete a urine pregnancy test at the Biodynamics Lab prior to X-ray, CT or MRI scans. The results of the pregnancy test will be documented by either the PI or Research Assistant and retained in a separate folder that is identified only by the participant's Study ID number.

Functional biomechanical outcomes will be measured at 6 months and 12 months using DSX at the Biodynamics Lab. Data will be obtained from the bilateral knees while the subjects perform a downhill running and a cutting maneuver task to simulate pivoting, each task will be repeated three times to ensure capture of movement. There will be at most 3 static standing trials before each movement tasks to image each knee. Participants will be tested within a biplane X-ray system throughout the study. Biplane radiographic images of each knee will be taken for 20 surgical patients, randomly assigned to ACL-R or ACL-R+EAT .

In the patient prep-room of the Biodynamics Lab, a member of the research team will place reflective markers throughout the body. Movement of the reflective markers will be tracked using conventional optical motion tracking equipment (Vicon MX).

Novel's pedar system will be used to measure pressure distribution under the foot for each participant during the dynamic movement trials. Each participant will be fitted with an elastic sensor insole (1.9 mm thickness) which will be connected to a data logging pack via cables. The cables will be secured around the participant's legs with velcro to minimize potential interference during the movement trials. The data logging pack will be fitted on a belt that will sit around the participants hip. The data logging pack will send data to the computer system via Bluetooth.

All trials will be performed on an instrumented treadmill that will collect ground reaction forces at 1000 Hz during each movement trial. This system contains two side-by side 30x180 cm belts. The belts are driven by independent (but synchronized) motor systems, and each belt/motor is configured on a rigid platform supported by multi-axis load cells. This configuration enables assessment of three-dimensional foot-ground reaction forces (vertical/ medial/lateral and anterior/posterior), applied torque and center-of-pressure location independently for each foot. The participants will perform some activities for the ankle on risers placed on the treadmill belt in order to image the ankle with the DSX machines. The treadmill belt will not move for the ankle trials, it will just be used to determine ground reaction forces.

The demographic questionnaire will then be completed and the PI, Research Assistant or Lab Manager will place the questionnaire into the folder containing de-identified participant information. This will include age, sex, height, weight and body mass index (BMI) along with standard anthropometric measurements used by our Vicon Nexus motion measurement system. Participants will aslo fill out the following questionnaires: IKDC subjective, KOOS, SAS97, VAS, Marx activity level, Lysohm Scale and VR-12.

ELIGIBILITY:
INCLUSION CRITERIA:

1. between age of 14-40
2. BMI between 18-35
3. have a contralateral healthy knee and within 12 months of grade 3 injury to the ipsilateral ACL
4. no greater than grade 2 injury to MCL or LCL and absence of PCL injury
5. articular cartilage injury grade 2 or lower
6. display a quantitative pivot shift test of >=3 mm lateral translation or >8 m/sec*2, or a side to side difference of 50% or greater
7. Use of a quad tendon graft or BTB graft

EXCLUSION CRITERIA:

* Subjects will have no other injury or disease that will interfere with knee function. Subjects will be of generally good health and will have decided to undergo ACL reconstruction surgery and agreed to participate in the study (following informed consent procedures).
* Potential candidates who do not intend to stay in the Pittsburgh area for a period of at least a year following surgery will be excluded.
* Pregnant females will be excluded. Urine pregnancy tests will be administered by the PI prior to research-related exposure to radiation (CT scan, Biodynamics Lab testing). If these radiation exposures occur on the same date, only one pregnancy test will be administered. If these radiation exposures occur on different dates, a pregnancy test will be administered each date.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2019-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change of joint kinematics | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  Outcome data includes: Joint contact path, functional joint space, anterior translation, varus-valgus rotation, and internal-external rotation will be obtained.
Change in IKDC subjective | Surgical Visit
  The international knee documentation committee's objective scale will be used to record the surgical procedure on the knee.
Demographic Questionnaire | Visit 1 (up to two weeks prior to surgery)
  This will include race, age, sex, height and weight.
Change in KOOS | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  The knee injury and Osteoarthritis Outcome Score is used to access the subjects view on the knee injury.
Change in VAS | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  This visual scale will be used by the subject to report the level of pain at the time of testing.
Change in Marx Activity Scale | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  This scale will be used by the subject to report level of activity in the past year.
Change in Lysohm Scale | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  This scale will be used by the subject to report how the knee problems have affected management of daily life.
Change in VR-12 | Visit 1 (up to 2 weeks prior to surgery) and Visit 2 (3-6 months after surgery)
  This scale will be used by the subject to measure health related to quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: William Anderst, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Biodynamics Lab, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiba D, Gale T, Nishida K, Suntaxi F, Lesniak BP, Fu FH, Anderst W, Musahl V. Lateral Extra-articular Tenodesis Contributes Little to Change In Vivo Kinematics After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Am J Sports Med. 2021 Jun;49(7):1803-1812. doi: 10.1177/03635465211003298. Epub 2021 Apr 19. PMID 33872056
- [Derived] Nishida K, Gale T, Chiba D, Suntaxi F, Lesniak B, Fu F, Anderst W, Musahl V. The effect of lateral extra-articular tenodesis on in vivo cartilage contact in combined anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2022 Jan;30(1):61-70. doi: 10.1007/s00167-021-06480-4. Epub 2021 Feb 12. PMID 33580345